CLINICAL TRIAL: NCT03572998
Title: Lymphatic Function in Patients Who Have Undergone Breast Cancer Treatment
Acronym: LYFE-B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 220493; 1-10-72-193-18 (Registry Identifier: De Videnskabsetiske Komitéer for Region Midtjylland)
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Secondary Lymphedema
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Case-control. Patients function as their own control since the treated arm will be compared with the non-treated arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer patients (Other): study subject
  Interventions: Drug: Indocyanine Green (ICG)

INTERVENTIONS:
Drug: Indocyanine Green (ICG) — Injection of ICG as a fluorophore for Near Infrared fluorescence Imaging (NIRF)

SUMMARY:
Protocol resume

Swelling of tissue due to excess fluid, called lymphedema, is a common side effect of breast cancer treatment that requires lifelong treatment but in what way the treatment of breast cancer affects the lymphatic vasculature is not yet fully understood.

The overall aim of this study is to examine the baseline lymphatic function and anatomy in women who have undergone and completed treatment for breast cancer.

Comparison will be made between:

* The treated arm and the untreated arm in the participant.
* The treated arm in patients who did not develop lymphedema and the treated arm in patients who did.

By using an emerging technique, Near Infrared fluorescence imaging (NIRF), and non-contrast MRI it is now possible to examine the link between breast cancer treatment and the development of lymphedema. This project will describe the impact of breast cancer treatment on contractile function and morphological changes of the lymphatic vasculature in the upper extremity in patients treated for breast cancer.

The study population will consist of 28 patients treated for breast cancer who simultaneously are enrolled in the Skagen 1 trial. The NIRF imaging and MRI will be performed after completion of breast cancer treatment and no later than half a year after completion treatment. All examinations will be made under similar conditions, on the same segment of lymphatic vasculature, in the same room and bed and with patients in the supine position. The estimated duration of each examination is approximately 3,5 hours.

Upon arrival participants will receive three injections of ICG distally on each arm, two on the dorsal side and one on the palmar side. Ten minutes after injection, the primary sequence of the lymphatic vessels will be recorded, allowing for calculation of frequency and velocity. Following, the pumping pressure of the lymphatic vessels will be estimated. After completion of the NIRF examination, an MRI scan of the upper body and extremities will be made, allowing for morphological evaluation of the lymphatic system in the region.

By studying the lymphatic vessels in these patients, data may elucidate the characteristics of the changes taking place and thus provide new insight for future studies and possibly future treatments and ways to prevent or reduce the development of edema.

DETAILED DESCRIPTION:
Aim:

The overall aim of this study is to examine the baseline lymphatic function and anatomy in women who have undergone and completed treatment for breast cancer.

Comparison will be made between:

* The treated arm and the untreated arm in the patient.
* The treated arm in patients who did not develop lymphedema and the treated arm in patients who did.

Introduction:

The lymphatic vasculature is distributed around the entire body where it pumps excess protein-rich fluid from the interstitial space back to the circulatory system. It does so partly by intrinsic contraction of lymphatic smooth muscle cells in the lymphatic vessel wall and partly by the forces applied to the lymphatic vessels by surrounding contracting muscles. Lymphatic valves in the vessels prevent backflow of the fluid. Lymphedema occurs when the lymphatic vasculature is unable to transport the lymphatic fluid out of an affected region. (1) There are two types of lymphedema. The first is idiopathic lymphedema and consist of lymphedema caused by genetic dysfunction or inherent anatomical abnormalities of the lymphatic vasculature. The second type is called acquired lymphedema and is due to external factors such as physical disruption, compression of lymphatic vessels, surgery or radiotherapy. (2) The commonest reason for lymphedema in the western world is cancer treatment. It is seen after treatment of several different cancer types such as gynecologic cancer, melanoma, genitourinary cancer, head and neck cancers and particularly breast cancer being the most frequent cancer type in women in Denmark. (3-7) More than one in five patients surviving breast cancer experience lymphedema, however, estimates range from 13-65%.(8, 9) Radiation therapy to the breast or to the axilla appears to increase the risk of lymphedema significantly. (10-12) These patients experience a large number of severe consequences, both physical and psychological, following development of lymphedema. These include decrease of physical strength, range-of-motion and sense in the upper extremities. An increased feeling of pain and heaviness is also experienced. Psychologically, these women experience anxiety, depression, sexual dysfunction, reduced body confidence and a lowering of general quality of life. (13-18) The current treatment of lymphedema consists primarily of complete decongestive treatment (CDT), which combines different treatment approaches such as bandaging, compression garments, manual lymphatic drainage, and exercise. Although the current treatment options can help patients with lymphedema significantly, the patients still have to undergo a lifelong treatment and cope with some of the complications previously mentioned. (19) In order to secure a foundation for the development of curative or preventive treatments of lymphedema developed due to breast cancer treatment, the impact of this oncological treatment on the function and anatomy of the lymphatic vessels has to be understood.

Design:

Study population:

The study population will consist of 28 patients treated for breast cancer who simultaneously are enrolled in the Skagen 1 trial. The NIRF imaging and MRI will be performed after completion of breast cancer treatment and no later than half a year after completed treatment.

Information to the patient:

All women being candidates for the Skagen 1 Trial will be invited to participate in this study by their oncologist. If the patient is interested contact information will be passed along to the principal investigator. He and the participant will make an agreement of place and time for the meeting to happen and the participant will be informed that she is requested to participate in a health scientific research project. The participant is encouraged to bring along an assessor to the information. The meeting takes place in a quiet and undisturbed room affiliated with the Department of Cardiothoracic and Vascular Surgery. Oral as well as written information of the study are given to the participant and the procedures, the risks and the gains of the study are carefully explained. If the patient is interested in participating she will be asked to give her written consent. The patient will be told that she should consider it before deciding and that her consent is not binding and can be withdrawn at any time should she wish to do so. The study will be performed no earlier than two weeks after the information is given. Therefore, they will have two weeks to consider whether to participate or not.

After the meeting the participant will be informed:

* If new information regarding risks, side effects or complications emerges.
* If any changes to the research design is made that affects the participant.
* If new information regarding the health status of the participant emerges unless she has asked to not be informed.
* Of the results obtained and their consequences regarding the participant in she wishes.
* If the project is cancelled and the reason why.

Study procedures:

By using a novel lymphatic imaging technique, the Near Infrared Fluorescence imaging (NIRF), and non-contrast MRI scans the function and the anatomy of the lymphatic vasculature can be visualized and analyzed. These two imaging techniques have been shown to be superior to other techniques in lymphedema imaging. (20) All examinations will be made under similar conditions, on the same segment of lymphatic vasculature, in the same room and bed and with patients in the supine position. The estimated duration of each examination is approximately 3,5 hours.

NIRF setup: This study will be using a custom-built setup previously used by the Department of Cardiothoracic and Vascular Surgery at Aarhus University Hospital (21, 22): A EM-CCD camera (C9100-13 Hamatsu, Japan), with a Navitar lens (25mm f 0.95) and 835±15nm band-pass filters on each side of the lens. The light source is a custom designed 785 nm 450 mW laser (PowerTechnology, Arkansas, US). A 780±28nm band-pass filter is placed in front of the laser to minimize light leakage. Indocyanine Green (ICG) will be used as a fluorophore, and a 0,1 mL injection of 0.025% ICG dissolved in saline, equivalent to a 25μg dose per injection, will be given prior to commensal of the study.

Research design:

Near Infrared Fluorescence Imaging: In this study, different tests will be made to measure lymphatic activity.

Frequency and velocity: Contraction frequency and package velocity will be examined and calculated using LabView. Contraction frequency will be defined as lymphatic contractions generated per minute, and contraction package velocity as the velocity by which the lymph is propelled forward following each contraction.

Pumping pressure: A highly accurate (±1mmHg) cuff system (Hokanson E20 rapid cuff inflator, Hokanson AG101 air source) will be positioned around the proximal antebrachium, after having manually emptied the lymph vessels proximally to the cuff. The cuff will then be inflated to 80 mmHg, and after every 5 minutes, the pressure will be lowered by 5 mmHg. Over time the pressure of the lymphatic vessels will exceed that of the cuff, and lymph will pass through, giving an estimate of the pressure within the lymphatic vessel. The cuff will be placed identically during both examinations.

Magnetic Resonance Imaging: MRI will be used to visualize the anatomy and the morphology of the lymphatic system.

MRI: The lymphatic anatomy of the neck, entire chest, abdomen, and arms will be imaged and investigated with a 3 T MRI system (Siemens Skyra; Siemens Medical, Germany). MRI will included a respiratory-gated (navigator) 3D fast spin-echo sequence with the following parameters: matrix = 448 × 448, voxel size = 0.9 × 0.9 × 0.8 mm3 FOV = 100 - 400 cm2, repletion time = 2830 ms, echo time = 649 ms, flip angle = 125˚. This sequence will be repeated sequentially for whole-body coverage using multiple phased-array coils, with each coil covering a different body region, without coil repositioning

Protocol:

Upon arrival participants will receive three injections of ICG distally on each arm, two on the dorsal side and one on the palmar side. Ten minutes after injection, the primary sequence of the lymphatic vessels will be recorded, allowing for calculation of frequency and velocity. Following, the pumping pressure of the lymphatic vessels will be estimated as described above. All NIRF sequences will be recorded of the same region of lymphatic vessels and on both arms. After completion of the NIRF examination, an MRI scan of the upper body and extremities will be made, allowing for morphological evaluation of the lymphatic system in the region.

Study drug:

Drugs used as a tool:

ICG (0.5mg/ml solution) will be injected intradermally distally on each arm, two on the dorsal side and one on the palmar side for a total dose of 180μg. The Danish Health and Medicines Authority have approved the use of ICG to visualize lymphatic vessels using near infrared fluorescence in this study (reference number: LMST-2012025009). ICG green was FDA approved in the 1950's and has safely been used in different clinical procedures (ophthalmology, neurosurgery, hepatology and cardiology) ever since. In comparison to doses used in these procedures, up to 2mg/kg, the dose administered in the investigator's study (180μg) is considered small. ICG associates with albumin and as soon as it reaches the blood stream it is taken up by the liver and secreted into the bile, resulting in a biological half-life of 2-4 minutes in the blood. The only "side-effect" seen is a 4-5 mm green discolouration of the skin at the injections sites, which will disappear in a couple of days.

Side-effects:

The possible side effects of ICG (ICG-pulsion, Nomeco A/S, Denmark) are severe allergic reaction, which occurs very rarely (affects fewer than one in every 10,000 patients) and local irritation of the skin.

Together with the symptoms of the allergic reaction, an increase of special white blood cells associated with allergic reactions can occur (hypereosinophilia).

The possibility of an allergic reaction is greater in patients with extremely serious kidney failure.

Study duration:

The study will start September 1st, 2018 and terminate August 31st, 2019.

Ethical concerns Aside from the ICG injections and the discomfort of being inside an MRI machine, no inconvenience will be applied to the participants. The participants will not benefit from this study themselves other than knowing that they could contribute with knowledge that might enable a possible future treatment. The gain of knowledge this study provides outweighs the discomfort the participants may experience.

The participants participate on a voluntary basis with informed consent that can be withdrawn at any time. The participant's integrity and privacy will be respected. The study is conducted in accordance with the Helsinki declaration and Danish law.

Compensation to volunteers There will be no compensation to the participants.

Publication Positive, negative and inconclusive results will be published in an international scientific journal.

Clinical Perspectives:

The physiology behind the development of edema in breast cancer patients undergoing treatment is still not clear, however, a possible part of the explanation could be a change in function and/or anatomy of the lymphatic vessels after breast cancer treatment.

So far, the treatment of lymphedema is unsatisfactory. It is often life long treatment and invalidating for the quality of the patients life. If a change can be shown further studies can clarify what part or parts of the treatments are responsible for the change. This could be done by including patients before the start of treatment and then examine the patients after surgery/chemotherapy and after radiotherapy subsequently.

By studying the lymphatic vessels in these patients, data may elucidate the characteristics of the changes taking place and thus provide new insight for future treatments and ways to prevent or reduce the development of edema.

ELIGIBILITY:
Inclusion Criteria:

* Women who are being enrolled in the Skagen 1 Trial. The inclusion criteria for the Skagen 1 Trial and therefore this study is as follows:

  * Woman ≥ 18 years who had radical operation for invasive breast cancer pT1-3, pN0-N3, M0 with either mastectomy or breast conservation. The patient can be included no matter the status of estrogen receptor, progesterone receptor, malignancy grade, HER2 status.
  * Axillary lymph node dissection of the axilla where the findings give indication for regional nodes radiation therapy to levels (I), II, III, IV, interpectoral nodes and the IMN.
  * Sentinel node biopsy documenting limited nodal disease without an indication for axillary lymph node dissection according to institutional, national or other trial guidelines.
  * The patient may be a candidate for boost to the tumour bed.
  * Adjuvant systemic therapy with chemotherapy, endocrine therapy and anti-HER2 treatment is accepted.
  * Neoadjuvant chemotherapy to downstage a cT3-cT4 or cN2-cN3 breast cancer is accepted if there is not an indication for a boost in the area of regional nodes after surgery.
  * Primary systemic therapy of an operable breast cancer is accepted.
  * If the patient is not treated with chemotherapy she must be randomised within 42 days from last surgery. If she has received chemotherapy she must be randomised within 4 weeks after the last series of chemotherapy.
  * Breast implants are accepted.
  * Connective tissue disease is allowed if the treating clinical/radiation oncologist finds radiation therapy indicated.
  * Postoperative infection and/or seroma giving indication for drainage during RT is accepted
  * Patient with previous non-breast malignancy is accepted if the patient has been without disease minimum 5 years, and the treating oncologist estimates a low risk of recurrence. Patients with the following diseases can be accepted despite less than 5 years disease free interval: carcinoma in situ cervicis, carcinoma in situ coli, melanoma in situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin.
  * Life expectancy minimum 10 years.

Exclusion Criteria:

* Previous breast cancer or DCIS of the breast.
* Bilateral breast cancer.
* The patient has an indication for boost to 1 or more regional nodes.
* Previous radiation therapy to the chest region.
* Pregnant or lactating.
* Conditions indicating that the patient cannot go through the radiation therapy or follow up, or a condition where the treating oncologist thinks the patient should not participate in the trial for example due to language problems.
* Known iodide allergy.
* Claustrophobia.
* Foreign objects of metal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Pumping pressure | during the 3.5 hours study
  The pumping pressure in the lymphatic vessels.
Velocity | during the 3.5 hours study
  The velocity of the lymphatic fluid
Frequency | during the 3.5 hours study
  the frequency of contraction of the lymphatic vessels
morphology | During the 60 minutes MRI scan
  The morphology of the lymphatic vessels

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Hjortdal, professor, Principal Investigator — Department of Cardiothoracic and Vascular Surgery
Locations (1):
- Aarhus University, Aarhus C, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided